CLINICAL TRIAL: NCT03363789
Title: A Prospective Clinical Trial Comparing the Efficacy of Brisement to Physical Therapy for the Treatment of Achilles Tendinosis
Brief Title: The Efficacy of Brisement Compared to Physical Therapy for the Treatment of Achilles Tendinosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Chiodo, Division Chief, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P002307
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will analyze the data as group 1 and 2, not knowing which group received what treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brisement (Active Comparator): Patients will receive a series of brisement injections for treatment of non insertional Achilles tendinosis.
  Interventions: Biological: Brisement injection
- Physical Therapy (Active Comparator): Patients will undergo physical therapy for treatment of non insertional Achilles tendinosis.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Biological: Brisement injection — An injection of Lidocaine into the tendon sheath to break up adhesions that could be causing the condition.
  Arms: Brisement
Procedure: Physical Therapy — Patients will receive a prescription for physical therapy.
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of ultrasound guided brisement, brisement without ultrasound guidance and standard conservative treatment in patients who have been diagnosed with Achilles tendinosis. We are asking you to take part in this research study because you are a patient of the Brigham Foot and Ankle Clinic who has been diagnosed with Achilles tendinosis. About 100 people will take part in this research study, all at Brigham and Women's Hospital (BWH).

To our knowledge, there has been very little research in the efficacy of the addition of briesment injections to standard, conservative treatment of Achilles tendinosis. We hope our results will show which method is the most effective conservative treatment for Achilles tendinosis. This information will help doctors make decisions in the future.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the study must have a diagnosis of Achilles tendinosis with at least 2 weeks of pain at the distal Achilles tendon which is typically worsened with activity. Only cases of non-insertional Achilles tendinosis (tendinosis occurring above the point of tendon insertion) will be included.

Exclusion Criteria:

* Patients with a prior Achilles tendon tear, chronic inflammatory disease, or history of posterior calf surgery will be excluded from the study. Additionally, patients with prior injuries or fractures to the ankle and hind foot (talus and calcaneus) requiring surgery will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
VISA - A | 3 months

SECONDARY OUTCOMES:
PROMIS | 6 weeks, 3 months, 6 months, 1 year
VAS Pain Scale | Weekly for 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiodo, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.